CLINICAL TRIAL: NCT04938817
Title: A Phase 1b/2 Study to Evaluate the Efficacy and Safety of Investigational Agents as Monotherapy or in Combination With Pembrolizumab for the Treatment of Participants With PD-1/L1-refractory Extensive-Stage Small Cell Lung Cancer in Need of Second-Line Therapy (KEYNOTE-B98)
Brief Title: Safety and Efficacy Study of Investigational Agents as Monotherapy or in Combination With Pembrolizumab (MK-3475) for the Treatment of Extensive-Stage Small Cell Lung Cancer (ES-SCLC) in Need of Second-Line Therapy (MK-3475-B98/KEYNOTE-B98)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-B98; MK-3475-B98 (Other: MSD); KEYNOTE-B98 (Other: MSD); 2023-507687-38-00 (Registry Identifier: EU CT); U1111-1296-5646 (Registry Identifier: UTN); 2020-005628-12 (EudraCT Number)
Record Dates: First submitted 2021-06-21; First posted 2021-06-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Programmed Cell Death Receptor 1 (PD-1); Programmed Cell Death Receptor Ligand 1 (PD-L1); Programmed Cell Death Receptor Ligand 2 (PD-L2); PD-1; PDL1; PD-L1; PD-L2
MeSH Terms: conditions — Small Cell Lung Carcinoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Coformulation Pembrolizumab/Quavonlimab (Experimental): Participants receive pembrolizumab/quavonlimab (coformulation of pembrolizumab 400 mg and quavonlimab 25 mg) administered by intravenous (IV) infusion once every 6 weeks (Q6W) for up to 18 infusions (up to approximately 2 years) or until progressive disease or discontinuation.
  Interventions: Biological: coformulation pembrolizumab/quavonlimab
- Coformulation Pembrolizumab/Quavonlimab + Lenvatinib (Experimental): Participants receive pembrolizumab/quavonlimab (coformulation of pembrolizumab 400 mg and quavonlimab 25 mg) PLUS lenvatinib 20 mg. Pembrolizumab/quavonlimab will be administered by intravenous (IV) infusion once every 6 weeks (Q6W) for up to 18 infusions (up to approximately 2 years) or until progressive disease or discontinuation. Lenvatinib will be administered orally once-daily (QD) until progressive disease or discontinuation.
  Interventions: Biological: coformulation pembrolizumab/quavonlimab; Drug: lenvatinib
- Coformulation Pembrolizumab/Quavonlimab + MK-4830 (Experimental): Participants receive pembrolizumab/quavonlimab (coformulation of pembrolizumab 400 mg and quavonlimab 25 mg) PLUS MK-4830 800 mg. Pembrolizumab/quavonlimab will be administered by intravenous (IV) infusion once every 6 weeks (Q6W) for up to 18 infusions (up to approximately 2 years) or until progressive disease or discontinuation. MK-4830 will be administered by IV infusion once every 3 weeks (Q3W) for up to 36 infusions (up to approximately 2 years) or until progressive disease or discontinuation.
  Interventions: Biological: coformulation pembrolizumab/quavonlimab; Biological: MK-4830
- Coformulation Favezelimab/Pembrolizumab (Experimental): Participants receive favezelimab/pembrolizumab (coformulation of favezelimab 800 mg and pembrolizumab 200 mg) administered by intravenous (IV) infusion once every 3 weeks (Q3W) for up to 36 infusions (up to approximately 2 years) or until progressive disease or discontinuation.
  Interventions: Biological: coformulation favezelimab/pembrolizumab
- R-DXd (Experimental): Participants receive 5.6 mg/kg R-DXd via IV infusion every three weeks (Q3W) until progressive disease or discontinuation.
  Interventions: Biological: R-DXd

INTERVENTIONS:
Biological: coformulation pembrolizumab/quavonlimab — Intravenous (IV) infusion
  Other Names: MK-1308A
  Arms: Coformulation Pembrolizumab/Quavonlimab; Coformulation Pembrolizumab/Quavonlimab + Lenvatinib; Coformulation Pembrolizumab/Quavonlimab + MK-4830
Drug: lenvatinib — Oral administration
  Other Names: LENVIMA®; KISPLYX®; MK-7902; E7080
  Arms: Coformulation Pembrolizumab/Quavonlimab + Lenvatinib
Biological: MK-4830 — IV infusion
  Arms: Coformulation Pembrolizumab/Quavonlimab + MK-4830
Biological: coformulation favezelimab/pembrolizumab — IV infusion
  Other Names: MK-4280A
  Arms: Coformulation Favezelimab/Pembrolizumab
Biological: R-DXd — IV Infusion
  Arms: R-DXd

SUMMARY:
This study is a rolling arm study of investigational agents as monotherapy or in combination with pembrolizumab in participants with anti-programmed cell death 1 (PD-1)/ programmed cell death ligand 1 (PD-L1) refractory ES-SCLC in need of second-line treatment. This study will have 2 parts: an initial safety lead-in to determine safety and tolerability for experimental combinations of investigational agents without an established recommended phase 2 dose (RP2D) followed by an efficacy evaluation.

Investigational agents will initiate directly in or be added to the efficacy evaluation after an initial evaluation of safety and tolerability of the investigational agent has been completed in a separate study or in the safety lead-in of this study. If an RP2D for a combination being evaluated in the safety lead-in is established from another study, then the efficacy evaluation may begin at the determined RP2D.

There will be no hypothesis testing in this study.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Arms A-E:

  * Has histologically or cytologically confirmed diagnosis of ES-SCLC in need of second-line therapy
  * Has progressed on or after treatment with an anti-programmed cell death 1 (PD-1)/ programmed cell death ligand 1 (PD-L1) monoclonal antibody (mAb) administered as part of first-line platinum-based systemic therapy for ES-SCLC
  * Has ES-SCLC defined as Stage IV (T any, N any, M1a/b/c) by the American Joint Committee on Cancer, Eighth Edition
  * Has received 1 prior line of systemic therapy for small cell lung cancer (SCLC)
  * If a woman of childbearing potential (WOCBP), participant must have a negative highly sensitive pregnancy test within 24 hours (for a urine test) or 72 hours (for a serum test) before the first dose of study treatment
  * Has measurable disease per RECIST 1.1 as assessed by local site investigator/radiology and verified by BICR
  * Has submitted an archival tumor tissue sample or newly obtained core, incisional, or excisional biopsy of a tumor lesion not previously irradiated
  * Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 assessed within 7 days before allocation/randomization
  * Participants who are Hepatitis B surface antigen (HBsAg) positive are eligible if they have received Hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load before randomization
  * Participants with history of Hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening
  * Has a predicted life expectancy of >3 months
* Arms A-D:

  * Male participants must be abstinent from heterosexual intercourse or agree to use contraception during treatment for at least 7 days after the last dose of lenvatinib. No contraception is required if the participant is receiving pembrolizumab, pembrolizumab/quavonlimab, MK-4830, or favezelimab/pembrolizumab
  * Female participants are not pregnant or breastfeeding and are not a WOCBP or if are a WOCBP, are abstinent from heterosexual intercourse or are using contraception during the intervention period and for at least 120 days after the last dose of pembrolizumab, pembrolizumab/quavonlimab, MK-4830, or favezelimab/pembrolizumab or 30 days after the last dose of lenvatinib, whichever occurs last
  * Female participants must abstain from breastfeeding during the intervention period and for at least 120 days after the last dose of pembrolizumab, pembrolizumab/quavonlimab, MK-4830, or favezelimab/pembrolizumab or 7 days after the last dose of lenvatinib, whichever occurs last
* Has adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 millimeters of mercury (mm Hg) with no change in antihypertensive medications within 1 week before allocation/randomization
* Arm E:

  * If capable of producing sperm, the participant agrees to refrain from donating sperm and abstain from penile-vaginal intercourse or use a penile/external condom when having penile-vaginal intercourse with a nonparticipant of childbearing potential who is not currently pregnant. The length of time required to continue contraception for the study intervention R-Dx-d is 120 days
  * If a person of childbearing potential (POCBP) must use a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, or if they adhere to penile-vaginal intercourse abstinence as their preferred and usual lifestyle (abstinent on a long-term and persistent basis), during the intervention period and for at least the time needed to eliminate the study intervention after the last dose of study intervention. In addition, the participant agrees not to donate eggs (ova, oocytes) to others or freeze/store eggs during this period for the purpose of reproduction. The length of time required to continue contraception for the study intervention R-Dx-d is 210 days

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Arms A-E:

  * Has received prior systemic anticancer therapy including investigational agents within 4 weeks before start of study treatment
  * Has received prior radiotherapy within 2 weeks of start of study treatment
  * Has received lung radiation therapy >30 Gray (Gy) within 6 months before the first dose of study treatment
  * Has received a live or live attenuated vaccine within 30 days before the first dose of study treatment
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with brain metastases may participate only if they satisfy all of the following: completed treatment (e.g., whole brain radiation treatment, stereotactic radiosurgery, or equivalent) ≥14 days before the first dose of study intervention; have no evidence of new or enlarging brain metastases confirmed by post-treatment repeat brain imaging (using the same modality) performed ≥4 weeks after pretreatment brain imaging; and are neurologically stable without the need for steroids for ≥7 days before the first dose of study intervention as per local site assessment. Participants with untreated brain metastases will be allowed if they are asymptomatic, the investigator determines there is no immediate CNS-specific treatment required, there is no significant surrounding edema, and the brain metastases are of 5 millimeter (mm) or less in size and 3 or less in number.
* Has a history of severe hypersensitivity reaction (≥Grade 3) to any study treatment and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years except replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid)
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Arms A-D:

  * Has had major surgery within 3 weeks before first dose of study treatment
  * Has a preexisting ≥Grade 3 gastrointestinal or non-gastrointestinal fistula
  * Has clinically significant cardiovascular disease or major arterial thromboembolic event within 12 months before first dose of study intervention, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability
  * Has active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks before the first dose of study treatment
  * Has gastrointestinal malabsorption or any other condition that might affect oral study intervention absorption
  * Has serious nonhealing wound, ulcer, or bone fracture within 28 days before the start of study treatment
  * Has any major hemorrhage or venous thromboembolic events within 3 months before the start of study treatment
  * Has a history of inflammatory bowel disease
  * Has a history of a gastrointestinal perforation within 6 months before the start of study treatment
  * Has a known history of, or active, neurologic paraneoplastic syndrome
  * Has received prior therapy with a receptor tyrosine kinase (RTK) inhibitor or anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), anti-immunoglobulin-like transcript (ILT)-4, or anti-lymphocyte-activation gene 3 (LAG-3) agents
  * Has received prior therapy with an anti-PD-1/L1 agent and was permanently discontinued from that treatment due to a treatment-related adverse event
  * Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
  * Has radiographic evidence of encasement or invasion of a major blood vessel, or of intratumoral cavitation
  * Has symptomatic ascites, pleural effusion, or pericardial effusion
  * Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study treatment
  * Has a known history of Human Immunodeficiency Virus (HIV) infection
  * Has concurrent active HBV or HCV
  * Has progressive disease as initial response to first-line systemic chemotherapy in combination with PD-1/L1 inhibitor for ES-SCLC
  * Has had an allogenic tissue/solid organ transplant
* Arm E:

  * Received prior treatment with a CDH6-targeted agent or an ADC that consists of an exatecan derivative that is a topoisomerase I inhibitor (eg, trastuzumab deruxtecan, datopotamab deruxtecan)
  * Has received an investigational agent or has used an investigational device within 4 weeks (or 5 half-lives, whichever is shorter) prior to study intervention administration
  * Has Chronic steroid treatment (>10 mg/day prednisone [or equivalent] per day), except for inhaled steroids for asthma or COPD, mineralocorticoids (e.g., fludrocortisone) for participants with orthostatic hypotension, topical steroids for mild skin conditions, low-dose supplemental corticosteroids for adrenocortical insufficiency, Premedication for treatment groups and/or premedication in case of any hypersensitivity, or intra-articular steroid injections
  * Is an HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2029-12-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-Limiting Toxicities (DLTs) | Up to 21 days in Cycle 1 (Cycle 1 = 21 days)
  DLTs = ≥1 of the following treatment-related toxicities: Grade (G)4 nonhematologic toxicity; G4 hematologic toxicity lasting >7 days OR G4 platelet count decreased OR G3 platelet count decreased if associated with bleeding; G3 nonhematologic toxicity including G3 fatigue (lasting >3 days), G3 diarrhea, nausea, vomiting lasting ≥72 hours, G3 rash ≥7 days despite treatment, G3 uncontrolled hypertension; G3/4 nonhematologic laboratory abnormality if requires medical intervention, hospitalization, or persists for >1 week; G 3/4 febrile neutropenia, alanine aminotransferase, aspartate aminotransferase and/or bilirubin increase; drug-induced liver injury meeting the Hy's law; G4 creatinine increase; G4 electrolyte abnormalities; treatment related adverse event causing study intervention discontinuation during the first 21 days or administration delay >14 days during the first 21 days; G5 toxicity. The number of participants with ≥1 DLTs in the safety lead-in phase will be presented.
Number of Participants Who Experience at Least One Adverse Event (AE) | Up to approximately 60 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experience at least one AE will be presented.
Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE) | Up to approximately 60 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinue study treatment due to an AE will be presented.
Objective Response Rate (ORR) Per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 60 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 that has been modified for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) Per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 60 months
  PFS is defined as the time from randomization to the first radiographic disease progression (PD) or death due to any cause, whichever occurs first. PD is defined as at least a 20% increase in the sum of diameters (SOD) of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. RECIST 1.1 has been modified for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ. PFS as assessed by blinded independent central review (BICR) will be presented.
Duration of Response (DOR) Per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 60 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions), DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters (SOD) of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. RECIST 1.1 has been modified for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ. DOR as assessed by Blinded Independent Central Review (BICR) will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (48):
- United States (12):
  - Banner MD Anderson Cancer Center ( Site 0152), Gilbert, Arizona
  - Northside Hospital-Northside Hospital Oncology Network ( Site 0156), Atlanta, Georgia
  - Parkview Research Center at Parkview Regional Medical Center ( Site 0180), Fort Wayne, Indiana
  - Baptist Health Lexington-Research ( Site 0158), Lexington, Kentucky
  - University of Kentucky Chandler Medical Center-Medical Oncology ( Site 0157), Lexington, Kentucky
  - MFSMC-HJWCI-Oncology Research ( Site 0178), Baltimore, Maryland
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists ( Site 0172), Omaha, Nebraska
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists ( Site 0179), Omaha, Nebraska
  - Cleveland Clinic-Taussig Cancer Center ( Site 0166), Cleveland, Ohio
  - UPMC Hillman Cancer Center ( Site 0177), Pittsburgh, Pennsylvania
  - St Francis Cancer Center-Research Office ( Site 0167), Greenville, South Carolina
  - Virginia Cancer Institute ( Site 0169), Richmond, Virginia
- Australia (4):
  - Westmead Hospital-Department of Medical Oncology ( Site 4004), Westmead, New South Wales
  - The Prince Charles Hospital-Oncology Clinical Trials ( Site 4003), Brisbane, Queensland
  - Monash Health-Oncology Research ( Site 4005), Clayton, Victoria
  - Hollywood Private Hospital-Medical Oncology ( Site 4001), Perth, Western Australia
- Austria (2):
  - Standort Penzing der Klinik Ottakring-Abteilung für Atemwegs-und Lungenkrankheiten ( Site 3101), Vienna
  - Klinik Floridsdorf-Abteilung für Innere Medizin und Pneumologie ( Site 3100), Vienna
- Canada (3):
  - Cross Cancer Institute ( Site 3004), Edmonton, Alberta
  - Princess Margaret Cancer Centre ( Site 3003), Toronto, Ontario
  - St. Marys Hospital Center ( Site 3000), Montreal, Quebec
- Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház-Onkologiai Kozpont ( Site 3800), Szolnok, Jász-Nagykun-Szolnok, Hungary
- Israel (5):
  - Rambam Health Care Campus-Oncology ( Site 3600), Haifa
  - Shaare Zedek Medical Center-Oncology ( Site 3602), Jerusalem
  - Meir Medical Center. ( Site 3601), Kfar Saba
  - Rabin Medical Center-Oncology ( Site 3604), Petah Tikva
  - Sheba Medical Center-ONCOLOGY ( Site 3603), Ramat Gan
- Italy (4):
  - Humanitas-U.O di Oncologia medica ed Ematologia ( Site 3301), Rozzano, Milano
  - ospedale le scotte-U.O.C. Immunoterapia Oncologica ( Site 3300), Siena, Tuscany
  - Ospedale San Raffaele-Oncologia Medica ( Site 3303), Milan
  - Istituto Europeo di Oncologia IRCCS-Divisione di Oncologia Toracica ( Site 3304), Milan
- Poland (2):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier ( Site 3900), Warsaw, Masovian Voivodeship
  - Warminsko-Mazurskie Centrum Chorob Płuc w Olsztynie ( Site 3903), Olsztyn, Warmian-Masurian Voivodeship
- Russia (6):
  - Krasnoyarsk Regional Oncology Dispensary, Named after Krizhanovsky ( Site 3708), Krasnoyarsk, Krasnoyarsk Krai
  - Saint-Petersburg City Clinical Oncology Dispensary-Department of chemotherapy ( Site 3702), Saint Petersburg, Leningradskaya Oblast'
  - GBUZ LOKB-Oncology department #1 ( Site 3701), Saint Petersburg, Sankt-Peterburg
  - GBUZ "SPb CRPCstmc(o)" ( Site 3705), Saint Petersburg, Sankt-Peterburg
  - N.N.Petrov Research Institute of Oncology-Department of Chemotherapy and Innovative Technologies ( Site 3703), Saint Petersburg, Sankt-Peterburg
  - Scientific research institution of oncology named after N.N. Petrov-Thoracic oncology ( Site 3704), Saint Petersburg
- South Korea (5):
  - Seoul National University Bundang Hospital-Medical Oncology ( Site 4104), Seongnam, Kyonggi-do
  - Chungbuk National University Hospital ( Site 4106), Cheongju-si, North Chungcheong
  - Seoul National University Hospital ( Site 4101), Seoul
  - Asan Medical Center-Lung Cancer Center ( Site 4103), Seoul
  - Samsung Medical Center ( Site 4100), Seoul
- Spain (3):
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals ( Site 3403), L'Hospitalet de Llobregat, Catalonia
  - Hospital Universitari Vall d'Hebron-Oncology ( Site 3401), Barcelona
  - Hospital Clinic de Barcelona ( Site 3404), Barcelona
- Cantonal Hospital St.Gallen-Oncology & Hematology ( Site 3502), Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26347&tenant=MT_MSD_9011